CLINICAL TRIAL: NCT02395588
Title: Improving Heart Failure Outcomes (IHO)
Brief Title: Improving Heart Failure Outcomes Rural
Acronym: IHO Rural
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Other Study IDs: HP-00055798
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Guideline based care: Prior to discharge. Survey data will include descriptive characteristics, depression, heart failure knowledge. After patient education is complete prior to discharge patients will complete a readiness for discharge scale and heart failure self-care survey.
  Phone call 48 hours after discharge. Discharge instructions will be reinforced.
  Phone call 7 days after discharge. Survey data will include self management, complications, and satisfaction care.
  Secondary data 30 days post discharge. The hospital electronic medical record system will be queried to determine if the patient has been readmitted within 30 days of discharge for heart failure or non-heart failure causes.
  Interventions: Other: Guideline based care

INTERVENTIONS:
Other: Guideline based care — Patient education using guideline based teaching guides

SUMMARY:
This study will test if standardized care helps patients feel better, if it can be implemented in rural hospitals, and find out which healthcare processes and outcomes are most important to heart failure patients.

DETAILED DESCRIPTION:
The aims of this research are to: 1) Conduct a quasi-experimental study of rural hospitals to test if guideline-based care (standardized patient education, making a post discharge appointment with the patient's provider and calling the patient at 48 hours to reinforce HF education) improves patient outcomes (better self-care, and lower readmissions at 7 and 30 days post discharge); 2) Identify hospital (staffing, practice environment, costs) and provider (evidence-based practices) characteristics associated with better implementation of heart failure patient care processes; and 3) Determine which healthcare processes and outcomes are most important to heart failure patients. A quasi-experimental study with mixed methods will be used. The sample consists of HF patients (N=40, 20 each hospital) and nurses who care for HF patients on study units (N=90, 45 each hospital) from 2 rural hospitals. Survey data will be collected from patients (baseline, discharge, 48 hours and 7 days post discharge) and nurses (baseline, during patient education, on patient discharge). Secondary data will be collected quarterly on nurse staffing and once for patient readmission within 30 days of discharge. Structured patient interviews will be conducted with 10 HF patients in person to determine which health care processes and outcomes are most important to them. Both patients and nurses will be engaged to inform study procedures and outcomes consistent with the tenants of patient-centered outcomes research.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital with a diagnosis of heart failure
* Age > 20
* Cognitively intact
* English speaking
* Plan for discharge to home, assisted living or intermediate care

Exclusion Criteria:

* Patients with planned discharge to sub-acute or nursing home facilities
* Patients enrolled in another research study to test interventions to improve heart failure knowledge, self-management or reduce readmission to the hospital within 30 days post discharge
* Patients that are cognitively impaired
* Patients that are transferred to another unit in the hospital, and will be discharged from that unit
* Patients who undergo or have a planned surgical intervention during their hospital stay

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to participating rural hospitals with a diagnosis of heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Self-management | 7 Days
  Self-care of Heart Failure Index

SECONDARY OUTCOMES:
Readmission | 7 and 30 days post discharge
  Readmission to the hospital (all cause and heart failure related)

CONTACTS AND LOCATIONS:
Overall Officials: Robin P Newhouse, PhD, RN, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - Riverside Shore Memorial Hospital, Nassawadox, Virginia
  - Riverside Tappahannock Hospital, Tappahannock, Virginia